CLINICAL TRIAL: NCT05889923
Title: Training and Evaluation of Ultrasound-Guided Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clear Guide Medical (Industry)
Collaborators: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UMiami 2021
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Learning Anesthesia Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- learning with the EDU (Experimental): Students will perform 5 ultrasound-guided regional anesthesia procedures on a phantom using the EDU which shows the student how to hold the needle and probe to hit the target.
  Interventions: Device: With EDU

INTERVENTIONS:
Device: With EDU — using the EDU to perform the procedure

SUMMARY:
38 certified registered nurse anesthetist (CRNA) students will learn 5 different ultrasound-guided regional anesthesia blocks both with and without a novel device, the EDU which gives the student help finding the right needle path.

DETAILED DESCRIPTION:
38 students enrolled in a course for ultrasound-guided nerve blocks will be participants in a study to evaluate the benefit of learning with ultrasound guidance. The EDU, a computer assisted guide for ultrasound interventions will be used for half the students for each of 5 nerve blocks/interventional procedures. Then the students will switch (crossover study) and perform the same interventions. Data will be recorded by dint of the tiny video cameras on the EDU and anonymized and evaluated.

ELIGIBILITY:
Inclusion Criteria: All CRNA students in Dr. Hauglum's class on ultrasound-guided nerve blocks -

Exclusion Criteria: Any CRNA students who drop Dr. Hauglum's class on ultrasound-guided nerve blocks

-

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Distance to target | Day 1
  how close did the student come to the instructor-specified target
number of redirects | Day 1
  how many times did the student withdraw the needle and start again

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No